CLINICAL TRIAL: NCT01356914
Title: Randomized, Double-Blind, Placebo-Controlled, 4-Way Crossover Study to Evaluate the Safety, Tolerability and Effect on Atrial Fibrillation Burden of BMS-914392 in Patients With Paroxysmal Atrial Fibrillation and Permanent Pacemaker
Brief Title: Pacemaker Holter Assessment of the Effect of BMS-914392 on Atrial Fibrillation Burden
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV203-010; 2010-022947-39 (EudraCT Number)
Record Dates: First submitted 2011-04-15; First posted 2011-05-20 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A: BMS-914392 (Experimental)
  Interventions: Drug: BMS-914392
- Treatment B: BMS-914392 (Experimental)
  Interventions: Drug: BMS-914392
- Treatment C: BMS-914392 (Experimental)
  Interventions: Drug: BMS-914392
- Treatment D: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-914392 — Tablets, Oral, 10 mg, Every Day (QD), 20 days
  Arms: Treatment A: BMS-914392
Drug: BMS-914392 — Tablets, Oral, 10 mg, Three Times Daily (TID), 20 days
  Arms: Treatment B: BMS-914392
Drug: BMS-914392 — Tablets, Oral, 20 mg, Three Times Daily (TID), 20 days
  Arms: Treatment C: BMS-914392
Drug: Placebo — Tablets, Oral, 0 mg, Three Times Daily (TID), 20 days
  Arms: Treatment D: Placebo

SUMMARY:
The purpose of the study is to determine whether treatment with BMS-914392 is safe, well tolerated and associated with a reduction of atrial fibrillation burden in patients with paroxysmal atrial fibrillation and permanent pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation (AF)
* Programmable dual chamber pacemaker with appropriate arrhythmia diagnostics.
* 1-50% AF burden on pacemaker interrogation at screening.
* Women of childbearing potential (WOCBP) and men must be using an acceptable method of contraception to avoid pregnancy.

Exclusion Criteria:

* Persistent or permanent AF.
* AF Burden <1% or > 50%.
* Current or history of neurological diseases and mental disorders.
* Ejection Fraction < 45%.
* Severe mitral or aortic valve dysfunction.
* TIA (Transient Ischemic Attack) within last 12 months.
* Acute coronary syndrome in the last 2 months.
* Previous AF ablation.
* Cardioversion in last 3 months.
* Current kidney or liver disease, or current cancer.
* History of neurological and mental disorders.
* Major surgery within 4 weeks of first dose (cardiac surgery within 4 months).
* Screening lab test results outside of allowed limits per protocol.
* QTcF > 450 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation Burden | At screening (baseline)
Atrial Fibrillation Burden | Prior to randomization to study drug
Atrial Fibrillation Burden | On Day 1 of each cross-over period
Atrial Fibrillation Burden | On Day 8 of each cross-over period
Atrial Fibrillation Burden | On Day 22 of each cross-over period

SECONDARY OUTCOMES:
Number of participants with adverse events and type of adverse events | At Day 1 of each cross-over period
Number of participants with adverse events and type of adverse events | At Day 8 of each cross-over period
Number of participants with adverse events and type of adverse events | At Day 22 of each cross-over period
Number of Atrial fibrillation (AF) episodes | At Day 1 of each cross-over period
Number of AF episodes | At Day 8 of each cross-over period
Number of AF episodes | At Day 22 of each cross-over period
Duration of AF episodes | At Day 1 of each cross-over period
Duration of AF episodes | At Day 8 of each cross-over period
Duration of AF episodes | At Day 22 of each cross-over period
Heart Rate | At Day 1 of each cross-over period
Heart Rate | At Day 8 of each cross-over period
Heart Rate | At Day 22 of each cross-over period
Severity of AF (SAF) scale score at the end of each study period | At Day 1 of each cross-over period
Severity of AF (SAF) scale score at the end of each study period | At Day 8 of each cross-over period
Severity of AF (SAF) scale score at the end of each study period | At Day 22 of each cross-over period
Electrocardiogram (ECG) intervals (PR, QRS, RR, QT, QTc) | At Day 1 of each cross-over period
Electrocardiogram (ECG) intervals (PR, QRS, RR, QT, QTc) | At Day 8 of each cross-over period
Electrocardiogram (ECG) intervals (PR, QRS, RR, QT, QTc) | At Day 22 of each cross-over period
BMS-914392 plasma concentrations and exposures during each study period | At Days 1, 8 and 22 of each cross-over period

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Eastbourne General Hospital, Eastbourne, United Kingdom

REFERENCES:
- [Derived] Podd SJ, Freemantle N, Furniss SS, Sulke N. First clinical trial of specific IKACh blocker shows no reduction in atrial fibrillation burden in patients with paroxysmal atrial fibrillation: pacemaker assessment of BMS 914392 in patients with paroxysmal atrial fibrillation. Europace. 2016 Mar;18(3):340-6. doi: 10.1093/europace/euv263. Epub 2015 Oct 12. PMID 26462707